CLINICAL TRIAL: NCT00017108
Title: Low Dose Chlorambucil Maintenance Vs. No Treatment Following High-Dose Chlorambucil Induction In Patients With Advanced B-Chronic Lymphocytic Leukemia. A Randomized Phase III Study Of The EORTC LG (CLL-3)
Brief Title: Chlorambucil in Treating Patients With Advanced Chronic Lymphocytic Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068650; EORTC-06992-CLL-3
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2004-06

CONDITIONS: Leukemia
Keywords: stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Chlorambucil; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Drug: chlorambucil
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known which chlorambucil regimen is more effective in treating advanced chronic lymphocytic leukemia.

PURPOSE: Randomized phase III trial to determine the effectiveness of different regimens of chlorambucil in treating patients who have advanced chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall and disease-related survival of patients with B-cell chronic lymphocytic leukemia treated with high-dose chlorambucil induction therapy with or without low-dose chlorambucil maintenance therapy.
* Compare the time to salvage treatment in these patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare the treatment-related mortality of these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, time to complete response (before 12 weeks vs after 12 weeks vs partial response), and cytopenia at diagnosis (Binet stage A+B vs C).

All patients receive induction therapy comprising high-dose oral chlorambucil daily. Treatment continues until achievement of complete response or a maximum of 24 weeks in the absence of disease progression or unacceptable toxicity.

Patients who respond to induction therapy are randomized to 1 of 2 treatment arms for maintenance therapy.

* Arm I: Patients receive low-dose oral chlorambucil twice a week. Therapy continues for up to 5 years in the absence of disease progression or unacceptable toxicity. If disease progression occurs, then patients may proceed to salvage therapy.
* Arm II: Patients receive no maintenance therapy. If disease progresses, patients receive induction therapy again. If disease does not respond to re-induction therapy, then patients may proceed to salvage therapy.
* Salvage therapy: Patients with progressive disease during maintenance therapy receive fludarabine IV daily and cyclophosphamide IV daily on days 1-3. Treatment repeats every 4 weeks for 3-6 courses.

Patients are followed monthly for 3 months, every 2 months for 6 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: Approximately 470 patients will be accrued for this study within 4.7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia

  * Co-expression of CD5/CD19 or CD5/CD20 positivity, dim sIg, and CD23 positivity
  * Previously untreated advanced disease defined as presence of at least 1 of the following:

    * Total tumor mass (TTM) score greater than 9
    * TTM doubling time less than 12 months
    * Bone marrow failure (platelet count less than 100,000/mm^3 and/or hemoglobin less than 10 g/dL)

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin less than 3 times upper limit of normal (ULN)
* Hepatitis B negative
* No active hepatitis C

Renal:

* Creatinine less than 3 times ULN OR
* Creatinine clearance greater than 0.5 times normal

Cardiovascular:

* No severe cardiovascular disease
* No arrhythmia requiring chronic treatment
* No New York Heart Association class III or IV congestive heart failure
* No symptomatic ischemic heart disease

Other:

* No uncontrolled systemic infection
* HIV negative
* No prior or concurrent uncontrolled malignancy
* No prior or concurrent central nervous system or psychiatric disorders requiring hospitalization
* No psychological, familial, sociological, or geographical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior steroid therapy for less than 2 weeks allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03

CONTACTS AND LOCATIONS:
Overall Officials: Branimir Jaksic, MD, PhD — University of Zagreb Medical School
Locations (13):
- Belgium (3):
  - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hopital de Jolimont, Haine-Saint-Paul
- University Hospital - Olomouc, Olomouc, Czechia
- County Hospital, Kaposvár, Hungary
- Italy (2):
  - Azienda Ospedaliera Papardo, Messina
  - Ospedale Sant' Eugenio, Rome
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - Leyenburg Ziekenhuis, The Hague
- Clinical Center Skopje, Skopje, North Macedonia
- Hospital Escolar San Joao, Porto, Portugal